CLINICAL TRIAL: NCT06776263
Title: Dysfunctional Breathing in Patients With Post COVID-19 Condition
Brief Title: Dysfunctional Breathing in Post COVID-19 Condition.
Acronym: DB-PCC
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Nygren-Bonnier, PhD, Karolinska Institutet
Other Study IDs: 2024-05930-01
Record Dates: First submitted 2025-01-13; First posted 2025-01-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Post COVID-19 Condition (PCC); Dysfunctional Breathing; Breathing Pattern Disorder; Post-Acute COVID-19 Syndrome
Keywords: Respiration; Dyspnea; Signs and Symptoms, Respiratory; Hyperventilation; Outcome Assessment, Health Care; Patient Outcome Assessment; Surveys and Questionnaires
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Respiratory Aspiration; Dyspnea; Signs and Symptoms, Respiratory; Hyperventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with post COVID-19 condition.: Patients with post COVID-19 condition and respiratory problems.

SUMMARY:
The goal of this observational study with a cross-sectional design is to investigate what signs, symptoms and assessment which can describe and explain dysfunctional breathing in patients with post COVID-19 condition. The main question aims to answer which measurements can identify and asses dysfunctional breathing in patients with post COVID-19 condition?

Participants for this study will be recruited from the ReCov cohort will be evaluated with diffrent measurments and questionnaires.

DETAILED DESCRIPTION:
The overall aim with the proposed research project is to describe and investigate the underlying mechanisms of dysfunctional breathing and the experience of living with dysfunctional breathing in patients with post-COVID-19 conditions. In addition, validate and evaluate which methods measure dysfunctional breathing regarding content validity, conceptual validity, test-retest reliability, and sensitivity to change for patients with post-COVID-19 conditions. Furthermore, to develop and evaluate an individually adapted intervention with the aim of normalizing the breathing pattern. In the next step, to evaluate the effects of an individually adapted intervention on physical and psychological function and health-related quality of life (HRQoL) in patients with post-COVID-19 conditions, as well as to describe the patients' experiences of rehabilitation.

Methods and planned studies This project is a part of a larger multi-disciplinary and multi-professional study, ReCOV, that takes a holistic perspective on the consequences of the disease. ReCOV is a three-armed project including patients, next of kin and staff (23). Patients have been followed up at the out-patient clinic for patients with PCC at Karolinska University Hospital (K).

The longitudinal observational study is about physical and psychological recovery, objectively measured physical activity and also an interview study of the patients' overall experiences of rehabilitation after COVID-19 both in the acute and long-term perspective. In total approximately 950 patients have accepted to be apart of ReCOV and to this proposed project patients will be recruited from this cohort but also from primary care. This research project will be performed in collaboration with Karolinska Institutet, Karolinska university Hospital (K), Sahlgrenska University Hospital (SH). University of Gothenburg and primary care in Region Stockholm.

Study 1: Dysfunctional breathing in patients with post COVID-19 condition?

Aim: To investigate what signs, symptoms and assessment which can describe and explain dysfunctional breathing in patients with post COVID-19 condition.

Design: Cross-sectional design

Participants: Patients (approximately n=200) for this study will be recruited from the ReCov cohort. All patients will be > 18 years old. Patients that state that they have persistent respiratory problems and abnormal clinical respiratory findings will be included. Patients will also be recruited from primary care if they have suspected dysfunctional breathing pattern (unable to breathe with a normal breathing pattern in standing). Exclusion Criteria: Not able to perform the measurements because of cognitive or physical impairments, ongoing intervention of breathing exercises.

Procedure and outcomes: All included patients will be evaluated for physical and psychological function, symptoms and HrQoL. The following measurements and questionnaires will be used:

Dependent variables (primary outcome):

Health-related Quality of Life (EQ-5D-5L), EQ VAS Breathing pattern by Respiratory Movement Measuring Instrument (RMMI)

Independent, confounding and possible moderating variables:

Inspiratory and expiratory muscle strength (MIP and MEP) (Micro-RPM) Chest mobility by thoracic expansion Six-minute walk to measure endurance (in meters) Spirometry Diaphragmatic ultrasound End tidal CO2 measured during exercise

Physical Activity level (Frändin/ Grimby) Nijmegen questionnaire (dysfunctional breathing) COPD Assessment Test (CAT), questionnaire of symptoms related to breathing and now commonly used for this group of patients Dyspnea (mMRC, Modified Medical Research Council, Dyspnea Scale and BORG CR10) Patient Health Questionnaire (PHQ-9) Generalized Anxiety Disorder 7-item scale (GAD-7) Breathing Pattern Assessment Tool (BPAT)

ELIGIBILITY:
Inclusion Criteria:

* Patients that state that they have persistent respiratory problems, have 2 or higher on mMRC scale or 23 and over on the Nijmegen scale will be included.

Exclusion Criteria:

* Not able to perform the measurements because of cognitive or physical impairments, ongoing intervention of breathing exercises.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (approximately n=200) for this study will be recruited from the ReCov cohort. All patients will be > 18 years old. Patients that state that they have persistent respiratory problems and abnormal clinical respiratory findings will be included. Patients will also be recruited from primary care if they have suspected dysfunctional breathing pattern (unable to breathe with a normal breathing pattern in standing)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Breathing pattern by Respiratory Movement Measuring Instrument (RMMI) and Health-related Quality of Life (EQ-5D-5L) | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Will be assesed in a supine position, using the RMMI. First, during 30 seconds of tidal volume breathing. Second, during 60 seconds of performing maximal breathing manoeuvres interspaced by tidal volume breathing and then during 60 seconds after performing activity that triggers dyspnea. The RMMI records bilateral changes in the anterior posterior diameter, including both upper and lower thoracic and abdominal movements.
  Health-related Quality of Life is measured with EuroQualityOf Life 5 dimensions questionnaire (EQ-5D-5L), which is an instrument that evaluates the generic quality of life. EQ-5D includes a descriptive system, which comprises 5 dimensions of health: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. A descriptive index-score between 0-1, higher score indicates higher HRQoL. EQ-5D also includes a visual analog scale (VAS), which records self-rated health status on a graduated (0-100) scale, with higher scores for higher HRQoL

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Maximal Inspiratory muscle strength (MIP) will be measured with Micro RPM in cmH2O
Maximal Expiratory Pressure ( MEP) | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Maximal expiratory muscle strength (MEP) will be measured with Micro-RPM in cm H20
Chest mobility | Assessment will be applied only once and takes about 5 minutes to be completed.
  Chest mobility will be measured with a tape measure at the xiphoid process and the 4th rib
Six-minute walk test (6MWT) | Assessment will be applied only once and takes about 15 minutes to be completed.
  Six-minute walk to measure endurance (in meters)
Spirometry | Assessment will be applied only once and takes about 30 minutes to be completed.
  Lung function test with forced vital capacity (FVC), forced expiratory flow in one second (FEV1), diffusion capacity (DLCO)
End tidal CO2 | Assessment will be applied only once and takes about 15 minutes to be completed.
  End tidal CO2 measured during exercise
Physical Activity level (Frändin/ Grimby) | Assessment will be applied only once and takes about 2 minutes to be completed.
  Measured with Frändin/Grimby activity scale, which is a self-assessment scale about current levels of physical activity, ranging from 1 to 6. The higher the score, the higher level of physical activity.
Nijmegen questionnaire (dysfunctional breathing) | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Dysfunctional breathing will be assessed with the Nijmegen questionnaire. The questionnaire consists of 16 items asking about the symptoms related to dysfunctional breathing.
  Participants will grade how often they suffered from each item on a five-point Likert scale, ranging from 0 to 4, in which 0 is never ,1 is rarely, 2 is sometimes , 3 is often , and 4 is very often. Total score ranging from 0 to 64. A score of 23 and over indicates dysfunctional breathing.
COPD Assessment Test (CAT) | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  COPD Assessment Test (CAT), questionnaire of symptoms related to breathing and now commonly used for this group of patients. COPD Total score ranging from 0 to 40, where a higher number indicates more symptoms
Dyspnea | Assessment will be applied only once and takes about 5 minutes to be completed.
  Dyspnea (mMRC, Modified Medical Research Council 0-4), Dyspnea Scale and BORG CR10).
  Modified Medical Research Council (mMRC), which is a self-rating tool to measure the degree of disability that breathlessness postures on daily physical activities on a scale from 0 to 4. 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a hill; 2, walks slower than people of same age on the level because of breathlessness; 3, stops for breath when walking at their own pace on the level; and 4, Breathless when washing or getting dressed.
  Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
Depression | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Depression will be assessed with the Patient Health Questionnaire (PHQ-9). PHQ-9 which contains 9 items. Total score ranges from 0 to 27. Higher score indicate more severe depression symptoms
Anxiety | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  Anxiety will be assessed with the Generalized Anxiety Disorder 7-item scale (GAD-7) which is a self assessment tool. Total score ranging from 0-21. Higher score indicates higher anxiety.
Breathing Pattern | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  The Brompton BPAT (BREATHING PATTERN ASSESSMENT TOOL) will be used. Assessment components include (i) evaluation of chest/abdominal wall movement, noise of (ii) inspiratory and (iii) expiratory flow, (iv) channel of inspiration and expiration, (v) signs of air hunger (yawning, sighing and deeper breaths), (vi) RR and (vii) rhythm. Each component is given a score from 0 to 2, based on features consistent with expected normal (0) versus that present in severe dysfunctional breathing (2), giving a total score of between 0 and 14. The BPAT is completed with a patient positioned, as per the standard assessment of resting breathing pattern (i.e. sat comfortably in a supported seat for at least 5 min) and takes approximately 1 min to collate.
Thickness of the diaphragm | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  The thickness of the diaphragm will be measured using ultrasound at end-inspiration and end-expiration and is presented in cm.
Movement of the diaphragm | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  The movement of the diaphragm at rest, at deep breathing and at sniff manuver will be measured using ultrasound and presented in cm.
Velocity of the diaphragm | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  The velocity of the diaphragm movment will be measured with ultra sound and presented as cm/s.
Thickening fraction of the diaphragm | Assessment will be applied only once and takes about 5-10 minutes to be completed.
  The thickening fraction of the diaphragm will be measured using ultrasound and is calculated using a formula, thickening fraction=(end-inspiration - end-expration)/ end-expiraton ×100%. Measurements are performed 3 times and the average value is calculated and presented.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm, Solna
  - Karolinska Institutet, Huddinge

REFERENCES:
- See also: Related Info — https://www.webofscience.com/wos/alldb/citation-report/e227494f-d858-4197-87bc-c8c4e0e33290-01378fb818